CLINICAL TRIAL: NCT03870776
Title: Double-blind,Controlled,Randomized Phase 2 Study of Efficacy,Safety,Pharmacokinetics& Pharmacodynamics of Daily Oral Administration of MAP4343 During 6 Weeks in Antidepressant Non-responders Patients Experiencing a Major Depressive Episode
Brief Title: RESIST : Administration of MAP4343 in Antidepressant Non-Responders Patients Experiencing a Major Depressive Episode
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mapreg (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAP4343 / OP103617.MAP
Record Dates: First submitted 2019-02-26; First posted 2019-03-12 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Depression
Keywords: Depression; Resistant depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: There are 3 groups :
  * Placebo group will receive placebo during 42 days with antidepressant treatment in add-on.
  * Dose 1 during 42 days with antidepressant treatment in add-on. Upon IDMC recommendation after the first futility analysis (IDMC#5 13-Jun-2022), Dose 1 was stopped from the 17-Jun-2022.
  * Dose 2 during 42 days with antidepressant treatment in add-on.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group A (Placebo Comparator): Patients will receive the placebo during 42 days.
  Interventions: Drug: Placebo
- MAP4343 group B (Experimental): Patients will receive daily dose 1 during 42 days.
  Interventions: Drug: MAP4343
- MAP4343 group C (Experimental): Patients will receive daily dose 2 during 42 days.
  Interventions: Drug: MAP4343

INTERVENTIONS:
Drug: MAP4343 — Daily oral administration of MAP4343
  Arms: MAP4343 group B; MAP4343 group C
Drug: Placebo — Daily oral administration of Placebo
  Arms: Placebo group A

SUMMARY:
The study is a phase II, double-blind, randomized, placebo controlled, parallel, multicentric study in 110 patients with drug resistant depression.

DETAILED DESCRIPTION:
This is a phase II, versus placebo, multicentre, double blind, randomized, parallel study in male or female patients with drug resistant depression.

This study targets the antidepressant non-responders' patients who have already experienced at least 2 antidepressant treatments with no success. It is estimated that about 2/3 of the patients treated with antidepressant drugs do not respond partially or completely to the actual conventional treatments (Selective Serotonin Reuptake Inhibitor and Serotonin and Norepinephrine Reuptake Inhibitor).

110 patients with drug resistant depression episode, aged 18 to 80 will be included in the study. They will be recruited from psychiatric consultations in the centers participating to the study.

ELIGIBILITY:
Inclusion Criteria:

1. TRD level from to 2 to 4 inclusive according to the Thase & Rush classification;
2. Patient experiencing a Major Depressive Episode (MDE) according to DSM-5 criteria. MDE can be isolated or recurrent. The diagnosis is based on Mini-International Neuropsychiatric Interview (MINI) test;
3. Patient who received a previous antidepressant treatment (AD-Y) in monotherapy with vortioxetine, duloxetine or venlafaxine) at optimized dosages during 6 weeks prior to randomization, associated or not to AD-potentiator (quetiapine), are eligible.
4. Hamilton Depression Rating Scale (HDRS) score > 21;
5. Clinical Global Impressions scale (CGI) ≥ 4;
6. Male or female patient, aged 18 to 80 years inclusive;
7. Females of childbearing potential/Sexually active males with partner of childbearing potential: commitment to consistently and correctly use an acceptable method of birth control (oral, transdermal, systemic or implant contraception birth control, intrauterine devices, diaphragm or condoms) for the duration of the trial and for 4 months after the last study drug administration; Females of non-childbearing potential: either surgically sterilized or at least 1 year postmenopausal (amenorrhea duration at least 12 months);
8. Negative pregnancy test at screening baseline;
9. Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive;
10. Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests, urinalysis, hormonology). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator;
11. Normal ECG recording on a 12-lead ECG at the screening visit:

    * 120 < PR < 210 ms
    * QRS < 120 ms
    * QTcF ≤ 430 ms for male and < 450 ms for female,
    * No sign of any trouble of sinusal automatism,
    * Or considered NCs by investigators;
12. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 minutes in supine position:

    * 95 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 140 mmHg,
    * 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
    * 50 bpm ≤ HR ≤ 80 bpm,
    * Or considered NCs by investigators;
13. Signing a written informed consent prior to selection;
14. Covered by Health Insurance System and/or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. MDE with mood congruent or not congruent psychotic characteristics;
2. Patient hospitalized following the procedures: Psychiatric care at the request of another person (soins psychiatriques à la demande d'un tiers) or Psychiatric care at the request of the state representative (soins psychiatriques sur décision du représentant de l'Etat);
3. Suicidal risk in the last month before randomization (C-SSRS: answer yes to the item 3 and/or answer yes to section suicidal behavior; MINI 5.00; suicidal risk section or item 3 of HDRS ≥ 3);
4. History of other psychiatric disorder than DME except global anxiety, social phobia, panic troubles that should be accepted. In particular, patients who experienced a depressive state in bipolar disorder 1 or 2, schizophrenic or schizoaffective disorder should not be included;
5. Presence or history of drug hypersensitivity, or certain allergic-prone condition diagnosed that could represent a risk factor for an allergic shock;
6. Presence or history of hypersensitivity to vortioxetine, duloxetine, venlafaxine or one of their excipients;
7. Any history or presence of severe hepatic insufficiency and/or of hepatic disease which could lead to hepatic insufficiency;
8. Patients who are pregnant or breastfeeding. Patients should not be enrolled if they plan to become pregnant during the time of study participation;
9. Any drug intake during the last month prior to the first administration except treatments for concomitant pathologies which are stable since at least 3 months; Benzodiazepine-type anxiolytics, hydroxyzine chlorhydrate, and add-on treatments are authorized within limits described in Section 5.3; For the previous drug intake, the investigator should consider the time needed to sufficiently eliminate a drug from body system, e.g. 5 half-lives of the drug;
10. Subjects who received MAOI in monotherapy right before the selection (as ttX);
11. General anesthesia within 3 months before administration;
12. Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months;
13. Positive HBs antigen or anti HCV antibody, or positive results for HIV 1 or 2 tests;
14. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant, calculated creatinine clearance ≤ 60 mL/min;
15. Blood donation (including in the frame of a clinical trial) within 2 months before administration;
16. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
17. Medical history which in the opinion of the investigator would make the patient unsuitable for participation in the study (including, but not limited, to patients with coronary insufficiency, thromboembolism diseases);
18. Exclusion period of a previous study;
19. No possibility of contact in case of emergency;
20. History or presence of drug or alcohol abuse (alcohol consumption > 40 g/day);
21. Administrative or legal supervision.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale score evolution between baseline and D43 | 43 days
  Assessment of HDRS score with 17 items with sides 0 to 2 or 0 to 4. The scores from 0 to 4 correspond respectively to symptoms: absent, doubtful or insignificant, light, moderate, important, those ranging from 0 to 2 to symptoms: absent, doubtful or slight, overt or severe. The total score consists of the addition of the individual scores.

SECONDARY OUTCOMES:
Efficacy of treatment assessed by psychopathological evaluations with Hamilton Depression Rating Scale | 43 days
  psychopathological evaluations at each study visit: Hamilton Depression Rating Scale (17 items with sides 0 to 2 or 0 to 4. The scores from 0 to 4 correspond respectively to symptoms: absent, doubtful or insignificant, light, moderate, important, those ranging from 0 to 2 to symptoms: absent, doubtful or slight, overt or severe. The total score consists of the addition of the individual scores)
Efficacy of treatment assessed by psychopathological evaluations with Montgomery and Asberg Depression rating Scale | 43 days
  psychopathological evaluations at each study visit:Montgomery and Asberg Depression rating Scale used to quatify the intensity of depressive symptomatology
Efficacy of treatment assessed by psychopathological evaluations with Brief Anxiety Scale | 43 days
  psychopathological evaluations at each study visit: Brief Anxiety Scale, a dimensional measure of generalized anxiety with 8 items
Efficacy of treatment assessed by psychopathological evaluations with Scale of Global Clinical Impressions | 43 days
  psychopathological evaluations at each study visit: Scale of Global Clinical Impressions which includes 2 items rated from 1 to 7 (first item is a measurement of the overall measurement of patient's condition; 2nd item evaluates the overall improvementof patient compared to his condition at the admission to the research
Efficacy of treatment assessed by psychopathological evaluations with Quick Inventory of Depressive Symptoms | 43 days
  psychopathological evaluations at each study visit: Quick Inventory of Depressive Symptoms is a questionnaire allowing the assessment of the degree of depression by the patient himself.
Efficacy of treatment assessed by psychopathological evaluations with General Assessment Functioning | 43 days
  psychopathological evaluations at each study visit: General Assessment Functioning. The score is ranged on a hypothetical continuum from 1, the value representing the sickest individual, to 90, a value representing an individual without or with very minimal symptoms and functioning satisfactorily in his social environment or his family. The scale is divided into 9 equal intervals ranging from 1 to 10, 11 to 20, 21 to 30, etc.
Pharmacokinetic assessments with observed maximum plasma concentration (Cmax); | 127 days
  Cmax for MAP4343 in plasma at each study visit.
Pharmacokinetic assessments with first time to reach Cmax (tmax); | 127 days
  tmax for MAP4343 in plasma at each study visit.
Pharmacokinetic assessments with elimination rate constant (Kel); | 127 days
  Kel for MAP4343 in plasma at each study visit.
Pharmacokinetic assessments with plasma elimination half-life (t1/2); | 127 days
  t1/2 for MAP4343 in plasma at each study visit
Pharmacokinetic assessments with plasma area under the plasma concentration-time curve from administration up to infinity with extrapolation of the terminal phase (AUCinf); | 127 days
  AUCinf for MAP4343 in plasma at each study visit
Pharmacokinetic assessments with percentage of extrapolated AUCinf (%AUCextra); | 127 days
  %AUCextra for MAP4343 in plasma at each study visit
Pharmacokinetic assessments with volumn of distribution (Vd/F); | 127 days
  Vd/F for MAP4343 in plasma at each study visit.
Pharmacokinetic assessments with Clearance (Cl/F); | 127 days
  Cl/F for MAP4343 in plasma at each study visit
Pharmacokinetic assessments with accumulation ratio (R); | 127 days
  R for MAP4343 in plasma at each study visit.
Safety parameters assessed by the number of adverse events (AE) | 127 days
  AE evaluation
Safety parameters assessed - Heart rate | 127 days
  Vital signs assessed by heart rate measurement (beats per minute)
Safety parameters assessed by blood pressure | 127 days
  Vital signs assessed by systolic and diastolic blood pressure measurement (mmHg)
Safety parameters assessed - 12-lead Electrocardiogramm | 127 days
  Heart Rate; Electrocardiogramm measure during 12 hours (12-lead ECG) : heart rate (beats per minute)
Safety parameters assessed - 12-lead ElectrocardiogrammPR; | 127 days
  Electrocardiogramm measure during 12 hours (12-lead ECG) : PR interval (milliseconds)
Safety parameters assessed -12-lead Electrocardiogramm : QT | 127 days
  Electrocardiogramm measure during 12 hours (12-lead ECG) : QT interval (milliseconds)
Safety parameters assessed - 12-lead Electrocardiogramm : QTc | 127 days
  Electrocardiogramm measure during 12 hours (12-lead ECG) : QTc with automatic correction (milliseconds)
Safety parameters assessed by hematology parameters : Haemoglobin | 127 days
  Laboratory exams : hematology parameters (Haemoglobin in g/L)
Safety parameters assessed by hematology parameters: Haematocrit | 127 days
  Laboratory exams : hematology parameters (Haematocrit in %)
Safety parameters assessed by hematology parameters: Red blood cells | 127 days
  Laboratory exams : hematology parameters (Red blood cells in Tera/L)
Safety parameters assessed by hematology parameters: White blood cells | 127 days
  Laboratory exams : hematology parameters (White blood cells in Giga/L)
Safety parameters assessed by hematology parameters:Neutrophils | 127 days
  Laboratory exams : hematology parameters (Neutrophils in Giga/L
Safety parameters assessed by hematology parameters: Eosinophils | 127 days
  Laboratory exams : hematology parameters (Eosinophils in Giga/L)
Safety parameters assessed by hematology parameters: Basophils | 127 days
  Laboratory exams : hematology parameters (Basophils in Giga/L)
Safety parameters assessed by hematology parameters: Lymphocytes | 127 days
  Laboratory exams : hematology parameters (Lymphocytes in Giga/L)
Safety parameters assessed by hematology parameters: Monocytes | 127 days
  Laboratory exams : hematology parameters (Monocytes in Giga/L)
Safety parameters assessed by hematology parameters: Platelets | 127 days
  Laboratory exams : hematology parameters (Platelets in Giga/L)
Safety parameters assessed by hematology parameters: Reticulocytes; | 127 days
  Laboratory exams : hematology parameters (Reticulocytes in Giga/L)
Safety parameters assessed by red blood cells indices | 127 days
  MCV; Red blood cells indices : MCV (in picograms)
  MCH; Red blood cells indices : MCH (in picograms)
  MCHC; Red blood cells indices : MCHC (in picograms)
Safety parameters assessed by hemostasis parameters | 127 days
  INR measurement; Laboratory exams : hemostasis parameters (INR)
  Prothrombin time; Laboratory exams : hemostasis parameters (Prothrombin time in seconds)
  APTT; Laboratory exams : hemostasis parameters (APTT in seconds)
  APTT reference; Laboratory exams : hemostasis parameters (APTT reference in seconds)
Safety parameters assessed by serology parameters | 127 days
  P24 antigen; Laboratory exams : serology (P24 antigen detection)
  HIV; Laboratory exams : serology (HIV 1/2 antibodies detection)
  HCV; Laboratory exams : serology (HCV antibodies detection)
  HBs; Laboratory exams : serology (HBs antigen detection)
Safety parameters assessed by biochemistry parameters : Glucose | 127 days
  Lab exams: biochem(Glucose in mmol/L)
Safety parameters assessed by biochemistry parameters: Creatinine | 127 days
  Lab exams: biochem( in μmol/L)
Safety parameters assessed by biochemistry parameters: SGOT/ASAT | 127 days
  Lab exams : biochem(in IU/L)
Safety parameters assessed by biochemistry parameters: SGOT/ALAT | 127 days
  Lab exams: biochem(in IU/L)
Safety parameters assessed by biochemistry parameters:GGT | 127 days
  Lab exams: biochem(IU/L)
Safety parameters assessed by biochemistry parameters: Alkalin phosphatase | 127 days
  Lab exams: biochem(IU/L)
Safety parameters assessed by biochemistry parameters: CPK | 127 days
  Lab exams: biochem(IU/L)
Safety parameters assessed by biochemistry parameters: Total bilirubin | 127 days
  Lab exams: biochem(μmol/L)
Safety parameters assessed by biochemistry parameters: Conjugated bilirubin | 127 days
  Lab exams: biochem(μmol/L)
Safety parameters assessed by biochemistry parameters: Uric Acid | 127 days
  Lab exams: biochem(μmol/L)
Safety parameters assessed by biochemistry parameters: Cholesterol | 127 days
  Lab exams: biochem(in mmol/L)
Safety parameters assessed by biochemistry parameters: Triglycerides | 127 days
  Lab exams: biochem(in mmol/L)
Safety parameters assessed by biochemistry parameters: Sodium | 127 days
  Lab exams: biochem(in mmol/L)
Safety parameters assessed by biochemistry parameters: Potassium | 127 days
  Lab exams: biochem(in mmol/L)
Safety parameters assessed by biochemistry parameters: Chlore | 127 days
  Lab exams: biochem( in mmol/L)
Safety parameters assessed by biochemistry parameters:Calcium | 127 days
  Lab exams: biochem(in mmol/L)
Safety parameters assessed by biochemistry parameters:Total protein | 127 days
  Lab exams: biochem(in g/L)
Safety parameters assessed by biochemistry parameters:Albumin | 127 days
  Lab exams: biochem(in g/L)
Safety parameters assessed by hormonology parameters | 127 days
  Laboratory exams : hormonology (Β-HCG)
Safety parameters assessed by weight measurement | 127 days
  Physical exams : weight measurement in kilograms
Safety parameters assessed by height measurement | 127 days
  Physical exams : height measurement in centimeters
Battery of cognitive tasks | 43 days
  Cognitive evaluation
Plasmatic quantification of inflammatory biomarkers concentration (CRPs) | 43 days
  Plasmatic quantification of concentration CRPs.
Plasmatic quantification of inflammatory biomarkers concentration (Interleukins1, 6 and 10) | 43 days
  Plasmatic quantification of concentration of Interleukins 1, 6 and 10
Blood quantification of gut microbiome | 43
  Metagenomic study of blood markers of gut mircrobiome

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle VILLEY, PhD, MBA, Study Director — Mapreg
Locations (10):
- France (10):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - Cabinet Médical Ambroise Paré, Élancourt
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Fontan 1, Lille
  - CHU Nantes, Nantes
  - APHP Hôpital La Pitié Salpétrière - Prinicipal investigator center, Paris
  - Hôpital Ste Anne, Paris
  - CHU Henri Laborit, Poitiers
  - CHRU Tours, Tours